CLINICAL TRIAL: NCT07300436
Title: A Randomized, Open-label, Single-dose, Crossover Bioequivalence Study of TJ101 Injection Before and After CMC Change Following Subcutaneous Injection in Healthy Adult Male Subjects in China
Brief Title: A Study of TJ101 Injection Before and After CMC Change Following Subcutaneous Injection in Healthy Adult Male Subjects in China
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TJ101001BE102
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Males in China

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A（T-R） (Experimental)
  Interventions: Drug: TJ101 injection Test Product; Drug: TJ101 injection Reference Product
- Group B（R-T） (Experimental)
  Interventions: Drug: TJ101 injection Test Product; Drug: TJ101 injection Reference Product

INTERVENTIONS:
Drug: TJ101 injection Test Product — 1.2 mg/kg, administered by subcutaneous injection in the abdomen,Once per cycle
Drug: TJ101 injection Reference Product — 1.2 mg/kg, administered by subcutaneous injection in the abdomen,Once per period

SUMMARY:
This is Single-center, randomized, open-label, single-dose, two-period crossover study design.

The goal is to preliminary evaluate the PK comparability of TJ101 injection before and after CMC change following a single subcutaneous injection of 1.2 mg/kg in healthy male subjects in China, and to assess whether the two formulations are bio equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥ 18 and ≤ 45 years;
* Body mass index (BMI): 19-28 kg/m2 (inclusive), weight 50-90 kg (inclusive), with BMI calculated as: BMI = weight (kg) / height2 (m2);
* Results of physical examination, vital signs, laboratory tests, 12-lead ECG, chest X-ray (posteroanterior view), and abdominal B-scan ultrasound are normal or clinically insignificant if abnormal;
* Fully understand the purpose and requirements of this study, voluntarily participate in the clinical study and sign the written informed consent form (ICF), and are able to complete the entire study process as required.

Exclusion Criteria:

* (Screening/Admission interview) Known history of allergy to the investigational product, any of its components, or related products; or a history of allergic diseases such as asthma; or allergic diathesis (e.g., known allergy to two or more substances);
* (Screening/Admission interview) A definite history of diseases of the central nervous, cardiovascular, digestive, respiratory, urinary, or hematological systems, or metabolic disorders, or potential underlying diseases that are judged by the investigator to be clinically significant; or other diseases that the investigator considers unsuitable for participation in a clinical study (e.g., history of mental illness);
* (Screening/Admission interview) History of severe infection, severe trauma, or major surgery within 6 months prior to screening;
* (Screening/Admission interview) History of blood donation, blood loss ≥ 400 mL, or blood transfusion (at least one of the above) within 3 months prior to screening; or plan to donate blood within 3 months after the end of the study;
* Positive test for any of the following infectious diseases: human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis C virus antibody, Treponema pallidum specific antibody, and syphilis specific antibody;
* (Screening/Admission interview + Networked screening) Participation in any clinical trial of a drug, vaccine, or medical device within 3 months before the first dose (except for those who only signed the ICF but did not receive any drug, vaccine, or device intervention), or participated more than 3 months ago but are still in the follow-up period of a clinical trial or within 5 half-lives of the investigational drug (whichever is longer) before screening;
* (Screening/Admission interview) Use of any prescription drugs within 4 weeks before the first dose [including but not limited to any drugs that alter hepatic enzyme activity (e.g., glucocorticoids, sex hormones, anticonvulsants, cyclosporine, etc.)], or use of any over-the-counter drugs (including but not limited to Chinese herbal medicines, compound Chinese herbal preparations, health supplements, etc.) or vitamin supplements within 2 weeks before the first dose;
* (Screening/Admission interview) Prior use of growth hormone drugs;
* Positive for anti-TJ101 anti-drug antibody sample at screening;
* (Screening/Admission interview) History of drug abuse;
* (Screening/Admission interview) Smoke an average of ≥5 cigarettes per day within 3 months prior to screening, or are unable to stop using any tobacco products during the entire study period;
* (Screening/Admission interview) Alcoholic within 3 months prior to screening, defined as weekly alcohol use of more than 14 units (1 unit equals 17.5 mL or 14 g of pure alcohol; alcohol content of different types of alcoholic beverages is indicated by volume ratio, 1 unit of alcohol is approximately equal to 35 mL of 50-proof liquor or 350 mL of 5% beer), or are unwilling to stop alcohol use or consumption of any alcohol-containing products during the study period;
* (Admission period) Positive alcohol breath test or positive urine multi-drug panel test;
* (Screening interview) Difficulty with venipuncture and/or intolerance to intravenous paracentesis/indwelling needle, or have a phobia of needles or blood;
* (Screening/Admission interview) Have plans for procreation or sperm donation from the first dose of the investigational product until 3 months after the last dose, and are unwilling to take reliable contraceptive measures;
* (Screening physical examination) Any condition on the abdomen, such as scars or tattoos, that the investigator judges would interfere with the injection or observation of local reactions at the injection site;
* Other conditions that the investigator considers unsuitable for inclusion in this clinical study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-01-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary PK endpoint: Cmax | 10 days after dosing
  Maximum Concentration
Primary PK endpoint: AUC0-inf | 10 days after dosing
  Area Under the Concentration-Time Curve from Time Zero to Infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided